CLINICAL TRIAL: NCT01628523
Title: Mechanical Ventilation in the Emergency Department: A Prospective Cross-Sectional Study
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Iowa (Other); Christiana Care Health Services (Other); University of Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 201205165
Record Dates: First submitted 2012-06-20; First posted 2012-06-26 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Respiratory Failure; Mechanical Ventilation; Acute Lung Injury
Keywords: Respiratory failure; Mechanical ventilation; Acute lung injury
MeSH Terms: conditions — Respiratory Insufficiency; Acute Lung Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All ED patients requiring mechanical ventilation
  Interventions: Other: For inclusion in the study, patients will have to require mechanical ventilation either via an endotracheal tube or tracheostomy tube.

INTERVENTIONS:
Other: For inclusion in the study, patients will have to require mechanical ventilation either via an endotracheal tube or tracheostomy tube. — Mechanical ventilation via an endotracheal tube or tracheostomy tube

SUMMARY:
Despite its life-saving potential, the mechanical ventilator has great potential to do harm. Despite years of research, the mortality in acute lung injury (ALI) remains very high. Treatment options after ALI onset are very limited, therefore prevention may be the best option. Unfortunately, the emergency department has not been studied with respect to mechanical ventilation practices, and its contribution to ALI is unknown. The investigators hypothesize that mechanical ventilation is frequently used in the ED and for a variety of reasons, and that ED mechanical ventilation has an effect on long term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Ventilation either via an endotracheal tube or tracheostomy

Exclusion Criteria:

* Non-invasive positive pressure ventilation;
* Death in the immediate post-intubation phase of care;
* Chronic ventilator-dependence, either at home or extended care facility.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to the emergency department requiring invasive mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Fuller, MD, Principal Investigator — Washington University School of Medicine in St. Louis
Locations (4):
- United States (4):
  - Christiana Care Health System, Newark, Delaware
  - University of Iowa College of Medicine, Iowa City, Iowa
  - Washington University School of Medicine, St Louis, Missouri
  - University of Cincinnati College of Medicine, Cincinnati, Ohio

REFERENCES:
- [Derived] Fuller BM, Mohr NM, Miller CN, Deitchman AR, Levine BJ, Castagno N, Hassebroek EC, Dhedhi A, Scott-Wittenborn N, Grace E, Lehew C, Kollef MH. Mechanical Ventilation and ARDS in the ED: A Multicenter, Observational, Prospective, Cross-sectional Study. Chest. 2015 Aug;148(2):365-374. doi: 10.1378/chest.14-2476. PMID 25742126

RESULTS

PARTICIPANT FLOW:
Groups:
- All ED Patients Requiring Mechanical Ventilation: Assessed for mechanical ventilation parameters, predictors of ARDS in the patients without ARDS in the ED (n=204), and outcome differences between all patients with ARDS (n=45) and those not progressing to ARDS (n= 174). These 45 patients includes the 15 patients with ARDS in the ED and the 30 participants with incident ARDS after ED admission.
Period: Overall Study
Arm/Group | All ED Patients Requiring Mechanical Ventilation
Started | 219
Completed | 219
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Cohort: Characteristics of mechanically ventilated ED patients
Arm/Group | Entire Cohort
Number analyzed (Participants) | 219
Age, Customized [Mean (Standard Deviation); unit: years]
  age | 55.6 (19.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 128
Race/Ethnicity, Customized [Number; unit: participants]
  white | 152
  black | 59
  other | 8

OUTCOME MEASURES:

1. Primary Outcome: To Further Characterize ED Mechanical Ventilation
Description: In a prospective cross-sectional study design, we will enroll all patients receiving mechanical ventilation in the ED over a one-month time frame.
Time Frame: 1 month
Population: Tidal volume used for the entire cohort
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Entire Cohort
Number analyzed (Participants) | 219
mL | 500 [450 to 520]

2. Secondary Outcome: The Incidence of ARDS in Mechanically Ventilated Emergency Department Patients, and Risk Factors Associated With Progression to ARDS
Description: Development of ARDS after admission to the hospital
Time Frame: 1 month
Measure: Number; unit: participants
Groups:
- ARDS After Admission: Among the patients without ARDS while in the ED, these patients were analyzed for ARDS incidence after admission
Arm/Group | ARDS After Admission
Number analyzed (Participants) | 204
participants | 30
Statistical Analysis 1: Comparison: ARDS After Admission; Test type: Superiority or Other; p < 0.05, Regression, Logistic; Odds Ratio (OR) = 1.08

ADVERSE EVENTS:
Time Frame: Patients were enrolled for a month and followed until death or hospital discharge.
Arm/Group | All ED Patients Requiring Mechanical Ventilation
All-Cause Mortality (participants affected / at risk) | 72/219
Serious Adverse Events (participants affected / at risk) | 0/219
Other Adverse Events (participants affected / at risk) | 0/219

LIMITATIONS AND CAVEATS:
This was an observational study, so only associations (and not causation) can be concluded from the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No